CLINICAL TRIAL: NCT05498480
Title: A Phase 1 Study of Relatlimab (Anti-LAG-3 Monoclonal Antibody) in Combination With Nivolumab (Anti-PD-1 Monoclonal Antibody) in Chinese Participants With Advanced Solid Tumors
Brief Title: Study of Relatlimab in Combination With Nivolumab in Chinese Participants
Acronym: RELATIVITY-111
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA224-111
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; Relatlimab; Nivolumab
MeSH Terms: interventions — relatlimab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: Relatlimab Dose 1 + Nivolumab (Experimental)
  Interventions: Biological: Relatlimab; Biological: Nivolumab
- Cohort 2: Relatlimab Dose 2 + Nivolumab (Experimental)
  Interventions: Biological: Relatlimab; Biological: Nivolumab

INTERVENTIONS:
Biological: Relatlimab — Specified dose on specified days
  Other Names: BMS-986016
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo

SUMMARY:
The purpose of this study is to evaluate the safety and drug levels of relatlimab combined with nivolumab in Chinese participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologic or cytological confirmation of an incurable solid malignancy that is advanced (metastatic and/or unresectable) except for participants with primary central nervous system (CNS) tumors.
* Participants must have received, and then progressed or been intolerant to at least 1 standard treatment regimen in the advanced or metastatic setting (immune check inhibitor-experienced or non-experienced population may be included), if such a therapy exists. Participants who refuse or are ineligible for standard therapy will be allowed to enroll provided their refusal/ineligibility is documented in medical records.
* Eastern Cooperative Oncology Group (ECOG) 0 to 1.

Exclusion Criteria:

* Participants with history of severe and/or life-threatening toxicity related to prior immune therapy (eg, anti-cytotoxic T-lymphocyte-associated protein 4 [anti-CTLA-4] or anti-programmed cell death protein 1 [anti-PD-1]/programmed death-ligand 1 [PD-L1] treatment or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (eg, hormone replacement after endocrinopathy).
* Participants with an active, known, or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Prior treatment with LAG-3 targeted agents.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 123 Weeks
Number of Participants with Immune-mediated Adverse Events (IMAEs) | Up to 123 Weeks
Number of Participants with Serious Adverse Events (SAEs) | Up to 123 Weeks
Number of Deaths | Up to 123 Weeks
Number of Participants with AEs Leading to Discontinuation | Up to 123 Weeks
Number of Participants with Dose-Limiting Toxicities (DLTs) | Up to 123 Weeks
Number of Participants with Clinical Laboratory Abnormalities | Up to 123 Weeks
Maximum Observed Plasma Concentration (Cmax) of Relatlimab | Up to 123 Weeks
Time of Maximum Observed Plasma Concentration (Tmax) of Relatlimab | Up to 123 Weeks
Trough-observed serum concentration (Ctrough) of Relatlimab | Up to 123 Weeks

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Investigator | Up to 123 Weeks
Disease Control Rate (DCR) per RECIST v1.1 by Investigator | Up to 123 Weeks
Duration of Response (DOR) per RECIST v1.1 by Investigator | Up to 123 Weeks
Best Overall Response (BOR) per RECIST v1.1 by Investigator | Up to 123 Weeks
Ctrough of Nivolumab | Up to 123 Weeks
Observed Serum Concentration at End of Infusion (Ceoi) of Nivolumab | Up to 123 Weeks
Percentage of Participants Positive for Anti-drug Antibodies (ADAs) to Relatlimab | Up to 123 Weeks
Percentage of Participants Positive for ADAs to Nivolumab | Up to 123 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com